CLINICAL TRIAL: NCT04161534
Title: KT Tape Vs Arm Sling for Pediatric Clavicle Fractures
Brief Title: KT Tape for Pediatric Clavicle Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Shawn Gilbert, Professor, Chief of Pediatric Orthopaedics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300004149
Record Dates: First submitted 2019-10-11; First posted 2019-11-13 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Clavicle Fracture
Keywords: arm sling; Kinesiology tape

STUDY DESIGN:
Intervention Model Description: Participants will be treated with an arm sling and will be randomized to kinesio tape (KT Tape) or no kinesio tape (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm Sling Group (Active Comparator)
  Interventions: Device: Arm Sling
- KT Tape Group (Experimental)
  Interventions: Device: KT Tape; Device: Arm Sling

INTERVENTIONS:
Device: KT Tape — in addition to an arm sling, KT Tape will be applied to stabilize the clavicle fracture, thereby decreasing motion and pain.
  Arms: KT Tape Group
Device: Arm Sling — An arm sling will be applied to stabilize the clavicle fracture, thereby decreasing motion and pain.

SUMMARY:
Clavicle fractures in children are mostly managed non-operatively since they have an overall high union rate (95%) and a "good" functional outcome following nonoperative treatment. However, the downside of such a conservative approach is that patients have to live with pain and disability until the fracture heals. To minimize this, fractures are usually immobilized with a sling.

There have been no studies looking at clavicle fractures treated with kinesiology (elastic) tape. No adverse effects (skin irritation, redness, etc.) are observed with the application of this tape. Elastic tape has previously been examined regarding muscular advantages rather than for healing fractures. Since this tape should immobilize fractures better than a sling, patients should experience less pain and disability associated with their fracture.

ELIGIBILITY:
Inclusion Criteria:

* Clavicle Fracture
* Injury date within 1 week of presentation

Exclusion Criteria:

* Underlying neuromuscular disorder (eg osteogenesis imperfecta)
* Inability or unwillingness to report pain score until healing

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Score | Twice daily for 3 weeks, and one additional time 6 weeks after the initial injnury
  Participants will rate their pain on a scale from 1 to 10

SECONDARY OUTCOMES:
Change in Answers to DASH Questionnaire | Once weekly for 3 weeks, followed by one additional time 6 weeks after the initial injury.
  Participants will complete the DASH questionnaire to assess disability they might be experiencing due to their fracture.
Change in Analgesic Use | Once daily for 3 weeks, and one additional time 6 weeks after the initial injnury
  Participants will provide the need for taking analgesics (name, dose, and frequency).

CONTACTS AND LOCATIONS:
Overall Officials: Shawn R Gilbert, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's Hospital of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ersen A, Atalar AC, Birisik F, Saglam Y, Demirhan M. Comparison of simple arm sling and figure of eight clavicular bandage for midshaft clavicular fractures: a randomised controlled study. Bone Joint J. 2015 Nov;97-B(11):1562-5. doi: 10.1302/0301-620X.97B11.35588. PMID 26530661
- [Background] Reynard F, Vuistiner P, Leger B, Konzelmann M. Immediate and short-term effects of kinesiotaping on muscular activity, mobility, strength and pain after rotator cuff surgery: a crossover clinical trial. BMC Musculoskelet Disord. 2018 Aug 22;19(1):305. doi: 10.1186/s12891-018-2169-5. PMID 30134883
- [Background] Kaya E, Zinnuroglu M, Tugcu I. Kinesio taping compared to physical therapy modalities for the treatment of shoulder impingement syndrome. Clin Rheumatol. 2011 Feb;30(2):201-7. doi: 10.1007/s10067-010-1475-6. Epub 2010 Apr 30. PMID 20443039